CLINICAL TRIAL: NCT03849469
Title: A Phase 1 Multiple-Dose Study to Evaluate the Safety and Tolerability of XmAb®22841 Monotherapy and in Combination With Pembrolizumab in Subjects With Selected Advanced Solid Tumors (DUET-4)
Brief Title: A Study of XmAb®22841 Monotherapy & in Combination w/ Pembrolizumab in Subjects w/ Selected Advanced Solid Tumors
Acronym: DUET-4
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xencor, Inc. (Industry)
Collaborators: ICON Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XmAb22841-01; DUET-4 (Other: Xencor, Inc.)
Record Dates: First submitted 2019-02-19; First posted 2019-02-21 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Melanoma; Cervical Carcinoma; Pancreatic Carcinoma; Triple Negative Breast Cancer; Hepatocellular Carcinoma; Urothelial Carcinoma; Squamous Cell Carcinoma of the Head and Neck; Nasopharyngeal Carcinoma; Renal Cell Carcinoma; Non-small Cell Lung Carcinoma; Small Cell Lung Carcinoma; Gastric or Gastroesophageal Junction Adenocarcinoma; Advanced or Metastatic Solid Tumors; Prostate Carcinoma; Epithelial Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Carcinoma; Intrahepatic Cholangiocarcinoma; Squamous Cell Anal Cancer; Squamous Cell Penile Carcinoma; Squamous Cell Vulvar Carcinoma; Colorectal Carcinoma; Endometrial Carcinoma
Keywords: DUET-4; Advanced solid tumors; Metastatic solid tumors; Melanoma; Cervical Cancer; Pancreatic Cancer; Triple Negative Breast Cancer; Hepatocellular/Liver Cancer; Urothelial Cancer; Renal Cell Cancer; Squamous Cell Carcinoma of the Head and Neck; Non-small Cell Lung Cancer; Small Cell Lung Cancer; Gastric Cancer; Gastroesophageal Junction Cancer; Lymphocyte-activation gene 3 (LAG3); Cytotoxic T-lymphocyte-associated protein 4 (CTLA4); Prostate Cancer; Nasopharyngeal carcinoma; Epithelial ovarian cancer; Fallopian tube cancer; Primary peritoneal carcinoma; Intrahepatic cholangiocarcinoma; Squamous Cell Anal Carcinoma; Squamous Cell Penile Carcinoma; Squamous Cell Vulvar Carcinoma; Colorectal Carcinoma; Endometrial Carcinoma
MeSH Terms: conditions — Melanoma; Uterine Cervical Neoplasms; Pancreatic Neoplasms; Triple Negative Breast Neoplasms; Carcinoma, Hepatocellular; Carcinoma, Transitional Cell; Squamous Cell Carcinoma of Head and Neck; Nasopharyngeal Carcinoma; Carcinoma, Renal Cell; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Prostatic Neoplasms; Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms; Cholangiocarcinoma; Anus Neoplasms; Colorectal Neoplasms; Endometrial Neoplasms; Liver Neoplasms; Stomach Neoplasms; Diabetes Mellitus, Insulin-Dependent, 12 | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Arm 1: XmAb®22841 Monotherapy
  Interventions: Biological: XmAb®22841
- Arm 2 (Experimental): Arm 2: Combination of XmAb®22841 and Pembrolizumab (Keytruda®)
  Interventions: Biological: XmAb®22841; Biological: Pembrolizumab (Keytruda®)

INTERVENTIONS:
Biological: XmAb®22841 — Monoclonal bispecific antibody
Biological: Pembrolizumab (Keytruda®) — FDA-approved humanized monoclonal antibody
  Arms: Arm 2

SUMMARY:
This is a Phase 1, multiple dose, ascending-dose escalation study and expansion study designed to define a maximum tolerated dose and/or recommended dose of XmAb22841 monotherapy and in combination with pembrolizumab; to assess safety, tolerability, pharmacokinetics, immunogenicity, and anti-tumor activity of XmAb22841 monotherapy and in combination with pembrolizumab in subjects with select advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

PART A (Dose Escalation Cohorts)

1. All subjects' cancer must have progressed after treatment with all available therapies that are known to confer clinical benefit, or are intolerant to treatment, or refuse standard treatment.
2. All subjects must have adequate archival tumor, or give consent to a fresh tumor biopsy.
3. Subjects have an ECOG performance status of 0-1.
4. Subjects in monotherapy and combination therapy cohorts must have histologically or cytologically confirmed advanced or metastatic solid tumors, including the following:

   1. Melanoma
   2. Cervical carcinoma
   3. Pancreatic carcinoma
   4. Breast carcinoma that is estrogen receptor, progesterone receptor, and Her2 negative (TNBC)
   5. Hepatocellular carcinoma
   6. Urothelial carcinoma
   7. Squamous cell carcinoma of the head and neck (HNSCC)
   8. Nasopharyngeal carcinoma (NPC)
   9. Renal cell carcinoma
   10. Colorectal carcinoma or endometrial carcinoma
   11. Small cell lung carcinoma or NSCLC
   12. Gastric or gastroesophageal junction adenocarcinoma
   13. Prostate adenocarcinoma
   14. Epithelial ovarian cancer, fallopian tube cancer, or primary peritoneal cancer
   15. Intrahepatic cholangiocarcinoma
5. Subjects in the combination cohorts in Part A with XmAb22841 and pembrolizumab may have an advanced solid tumor that either:

   * has progressed after treatment with all available therapies that are known to confer clinical benefit, or is intolerant or has refused standard treatment (as for the XmAb22841 monotherapy cohorts), or
   * is of a tumor type for which pembrolizumab is an approved indication and has not previously been treated with an agent targeting PD1 or PDL1.

PART B (Dose Expansion Cohorts)

XmAb22841 Single Agent Cohort

1. Must have histologically or cytologically confirmed advanced or metastatic solid tumor that has progressed after treatment with all available therapies that are known to confer clinical benefit, or are intolerant to treatment, or refuse standard treatment. Eligible tumor types include the following:

1. Anti-PD1 refractory melanoma (or any uveal melanoma)
2. Anti-PD1 refractory NSCLC
3. Anti-PD1 refractory renal cell carcinoma (with clear cell component)
4. Anti-PD1 refractory urothelial carcinoma
5. Head and neck squamous cell carcinoma
6. Hepatocellular carcinoma
7. Gastric adenocarcinoma
8. Cervical carcinoma
9. Breast carcinoma that is estrogen receptor, progesterone receptor, and HER2 negative (TNBC)
10. Epithelial ovarian cancer
11. Nasopharyngeal carcinoma
12. Squamous cell anal carcinoma
13. Squamous cell penile carcinoma
14. Squamous cell vulvar carcinoma

XmAb22841 + Pembrolizumab Cohorts

1. Anti-PD-1 refractory melanoma (excluding uveal melanoma)
2. Anti-PD-1 naïve melanoma (excluding uveal melanoma)
3. Anti-PD-1 refractory NSCLC
4. Anti-PD1 naïve NSCLC

   a. Must be PD-L1 high (TPS ≥ 50%), with no EGFR or ALK aberrations
5. Anti-PD1 naïve urothelial carcinoma

   1. Must be PDL1 positive (CPS of ≥ 10), or ineligible for any platinum-containing chemotherapy regardless of PDL1 status; or
   2. Had disease progression within 12 months of neoadjuvant or adjuvant treatment with platinum-containing chemotherapy

Exclusion Criteria:

1. Prior treatment with an investigational anti-LAG3 therapy.
2. Treatment with any CTLA4 antibody within 16 weeks of the start of study drug for Cohorts 1M, 2M, 3M, 1P, and 2P; within 8 weeks for Cohorts 4M, 5M, 3P, 4P and 4Pi; and within 3 weeks for Cohorts 6M, 7Mi, 7M, 5P, and 6P.
3. Systemic antineoplastic therapy, unconjugated antibody therapy within 4 weeks of the first dose of study treatment; or radiotherapy within 2 weeks of the first dose of study treatment; or small molecule kinase inhibitors within 6 elimination half-lives of the first dose of study treatment.
4. Have received prior therapy with an anti-PD1, anti-PDL1, or anti PDL2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA4, OX 40, CD137) AND were permanently discontinued from that treatment due to an irAE.
5. Failure to recover from any irAE from prior cancer therapy to Grade ≤ 1.
6. Failure to recover from any other toxicity (other than immune-related toxicity) related to previous anticancer treatment to Grade ≤ 2.
7. Active known or suspected autoimmune disease (except that subjects are permitted to enroll if they have vitiligo; type 1 diabetes mellitus; residual hypothyroidism due to an autoimmune condition that is treatable with hormone replacement therapy only; psoriasis, atopic dermatitis, or another autoimmune skin condition that is managed without systemic therapy; or arthritis that is managed without systemic therapy beyond oral acetaminophen and non-steroidal anti-inflammatory drugs).
8. Receipt of an organ allograft.
9. Treatment with antibiotics within 14 days prior to first dose of study drug.
10. Participants with known HIV.
11. Participants with known chronic hepatitis B virus (HBV) infection treated for less than 3 months prior to study enrollment and/or with a detectable HBV viral load; or hepatitis C virus (HCV) infection that has been treated for less than 4 weeks prior to study enrollment and/or with a detectable HCV viral load; or active HBV/HCV coinfection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2023-02-16 (Actual); Study Completion 2023-02-16 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability profile of XmAb22841 assessed by rates of treatment-related adverse events (AEs), graded by CTCAE v4.03. | 56 Days
  Rates of treatment-related adverse events (AEs), graded by CTCAE v4.03, and additionally categorized as either immune-related or non-immune AEs.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Thompson, MD, PhD, Study Director — Xencor, Inc.
Locations (28):
- United States (28):
  - UCSD Medical Center - Encinitas, Encinitas, California
  - Koman Family Outpatient Pavilion, La Jolla, California
  - UC San Diego Medical Center - La Jolla (Jacobs Medical Center / Thornton Pavilion), La Jolla, California
  - UCSD Altman Clinical and Translational Research Institute Building (ACTRI), La Jolla, California
  - UCSD Perlman Medical Offices, La Jolla, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - UCLA Hematology & Oncology Clinic, Los Angeles, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - UCSD Rancho Bernardo Medical Office, San Diego, California
  - UCSD Medical Center - Vista, Vista, California
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Brigham and Women's Health Care Center, Chestnut Hill, Chestnut Hill, Massachusetts
  - University of Michigan Medical School, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Karmanos Cancer Institute Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Laura & Isaac Perlmutter Cancer Center at NYU Langone Health, New York, New York
  - NYU Langone Medical Center (Tisch Hospital), New York, New York
  - Columbia University Medical Center, New York, New York
  - Hospital of the University of Pennsylvania - Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - UPMC Shadyside Hospital, Pittsburgh, Pennsylvania
  - Mary Crowley Cancer Research - Medical City, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Utah, Huntsman Cancer Institute, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wong RL, Yu EY. Refining Immuno-Oncology Approaches in Metastatic Prostate Cancer: Transcending Current Limitations. Curr Treat Options Oncol. 2021 Jan 12;22(2):13. doi: 10.1007/s11864-020-00808-x. PMID 33433743